CLINICAL TRIAL: NCT00999713
Title: A Phase 3 Trial of Calfactant for ALI in Pediatric Leukemia and HSCT Patients
Brief Title: CALIPSO: Calfactant for Acute Lung Injury in Pediatric Stem Cell Transplant and Oncology Patients
Acronym: CALIPSO
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Neal Thomas, Neal J. Thomas, MD, Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Penn State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01FD003410-01 (FDA); R01FD003410-01A1 (FDA)
Record Dates: First submitted 2009-10-18; First posted 2009-10-22 (Estimated); Results first posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-02

CONDITIONS: Acute Lung Injury
Keywords: Acute Lung Injury; Cancer; Pediatrics
MeSH Terms: conditions — Acute Lung Injury; Neoplasms | interventions — calfactant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calfactant (Experimental): Endotracheal calfactant administration
  Interventions: Drug: Calfactant
- Placebo (air) (Placebo Comparator): Endotracheal air administration
  Interventions: Other: Air placebo

INTERVENTIONS:
Drug: Calfactant — Endotracheal calfactant, up to 3 doses if subject qualifies
  Arms: Calfactant
Other: Air placebo — Endotracheal air administration
  Arms: Placebo (air)

SUMMARY:
Acute lung injury (ALI) is a common, life-threatening complication among pediatric leukemia and lymphoma and hematopoietic stem cell transplant (HSCT) recipients. Although these children represent a relatively small and unique patient population, they account for the largest proportion of deaths of all pediatric diseases. The long-term goal of this project is to improve outcomes among these patients. Recently, the intratracheal administration of calfactant has resulted in decreased mortality among children with ALI including promising results among children with cancer and following HSCT. Consequently, the primary specific aim of this study is to assess the effect of calfactant on intensive care (PICU) survival among pediatric leukemia and lymphoma and HSCT patients with ALI. Secondary aims include assessment of the effect of calfactant on oxygenation and on the length of mechanical ventilation, PICU stay, and hospital stay. Calfactant therapy has been found to be of benefit in acute lung injury in the overall pediatric population by improving oxygenation and decreasing mortality. These findings, in conjunction with recent subgroup analysis in which calfactant therapy appeared to improve outcomes in immunocompromised children provide the rationale for assessing calfactant therapy in this patient population.

Funding Source - FDA Office of Orphan Products Development (OOPD)

ELIGIBILITY:
Inclusion Criteria:

1. Patients must meet criteria for acute lung injury

   * Intubated, mechanically ventilated, with respiratory failure secondary to diffuse, bilateral parenchymal lung disease (as judged by chest x-ray).
   * Oxygenation index (OI) > 13, but < 37, for two consecutive blood gases which should be separated by at least one hour within 48 hours of the initiation of mechanical ventilation.
   * Arterial catheter placement
   * Parental informed consent
2. Patients must have a diagnosis of leukemia/lymphoma undergoing active treatment or following HSCT for any indication. Leukemia/lymphoma will be defined according to the National Cancer Institute Surveillance Epidemiology and End Results Collaborative Staging Manual including those conditions defined as borderline such as myelodysplastic syndromes. All forms of HSCT will be eligible, allogeneic as well as autologous.

Exclusion Criteria:

1. Clinical diagnosis of congestive heart failure and/or pulmonary capillary wedge pressure >15 mmHg, or uncorrected congenital heart disease.
2. Glasgow Coma Score < 8 (prior to respiratory failure).
3. Pre-existing limitations on care options, (Do Not Attempt Resuscitation Orders, etc).
4. Patients with impending death from another disease.
5. Patients moribund or with other organ failure at possible randomization:

   * hypotension unresponsive to treatment (mean BP < 60 or < 5th % for age),
   * persistent cardiac tachyarrhythmia >150/minute, or persistent bradyarrythmia < 50/minute, or age appropriate criteria for younger children,
   * metabolic acidosis > - 10 milliequivalent (mEq)/L for more than 2 hours,
   * persistent arterial oxygen desaturation, arterial partial pressure of oxygen (PaO2) < 50 or oxygen saturation (SaO2) saturation < 80%,
   * hyperkalemia, serum K+ > 6.5 plus widening of QRS complex on EKG (QRS complex corresponds to the depolarization of the right and left ventricles of the heart).

Ages: 18 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2010-06; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal J Thomas, MD, MSc, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center; Robert F Tamburro, MD, MSc, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (16):
- United States (15):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Riley Children's Hospital, Indianapolis, Indiana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical Center, New York, New York
  - Maria Fareri Children's Hospital, Valhalla, New York
  - Rainbow Babies Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Hospital Sainte Justine, Montreal, Quebec, Canada

REFERENCES:
- [Background] Tamburro RF, Thomas NJ, Pon S, Jacobs BR, Dicarlo JV, Markovitz BP, Jefferson LS, Willson DF; Pediatric Acute Lung Injury and Sepsis Investigators (PALISI) Network. Post hoc analysis of calfactant use in immunocompromised children with acute lung injury: Impact and feasibility of further clinical trials. Pediatr Crit Care Med. 2008 Sep;9(5):459-64. doi: 10.1097/PCC.0b013e3181849bec. PMID 18679142
- [Background] Willson DF, Thomas NJ, Markovitz BP, Bauman LA, DiCarlo JV, Pon S, Jacobs BR, Jefferson LS, Conaway MR, Egan EA; Pediatric Acute Lung Injury and Sepsis Investigators. Effect of exogenous surfactant (calfactant) in pediatric acute lung injury: a randomized controlled trial. JAMA. 2005 Jan 26;293(4):470-6. doi: 10.1001/jama.293.4.470. PMID 15671432

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Calfactant | Placebo (Air)
Started | 26 | 17
Completed | 24 | 17
Not Completed | 2 | 0
Not completed — Physician Decision | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Calfactant | Placebo (Air) | Total
Number analyzed (Participants) | 26 | 17 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 16 | 39
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 5 | 15
  Male | 16 | 12 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 15 | 8 | 23
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 16 | 14 | 30
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Canada | 0 | 1 | 1
  United States | 26 | 16 | 42

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality at the Time of Pediatric Intensive Care Unit (PICU) Discharge
Description: Overall mortality rate from admission to PICU discharge
Time Frame: Admission to PICU discharge, up to 120 days
Measure: Count of Participants; unit: Participants
Arm/Group | Calfactant | Placebo (Air)
Number analyzed (Participants) | 26 | 17
Participants | 15 | 6

2. Secondary Outcome: Ventilator Free Days (VFDs)
Description: Number of days the patient is alive and off of the ventilator
Time Frame: 60 days after study enrollment
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Calfactant | Placebo (Air)
Number analyzed (Participants) | 26 | 17
Days | 0 [0 to 21.02] | 5.40 [0 to 17.44]

3. Secondary Outcome: Total Duration of Stay Required
Description: Length of stay (LOS) ,measured in days, from admission to PICU discharge and admission to hospital discharge.
Time Frame: Admission to discharge, up to 120 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Calfactant | Placebo (Air)
Number analyzed (Participants) | 26 | 17
days
  LOS from admission to PICU discharge | 15.5 [8 to 29.5] | 21 [12.5 to 39.5]
  LOS from admission to hospital discharge | 34.5 [17.5 to 95.5] | 65 [21 to 107.5]

4. Secondary Outcome: Change in Oxygenation: First Intervention
Description: The Oxygenation Index after the first intervention is calculated as the fraction of inspired oxygen, in percent, times the mean airway pressure, in mmHg, divided by the partial pressure of oxygen in arterial blood, in mmHg. Lower values are better.
Time Frame: 48 hours after enrollment, up to 12 hours after each intervention
Population: Total number of subjects analyzed at each measurement fluctuates due to arterial blood gas testing not being ordered at the appropriate time (i.e., subjects missing a test at a specific time point since the frequency of these tests in this study are not standard of care).
Measure: Geometric Mean (95% Confidence Interval); unit: index number
Arm/Group | Calfactant | Placebo (Air)
Number analyzed (Participants) | 24 | 17
index number
  First Intervention: Hour 0: number analyzed (Participants) | 22 | 16
  First Intervention: Hour 0 | 18.30178397 [14.8899734 to 22.49535894] | 20.59720208 [16.21205422 to 26.16847488]
  First Intervention: Hour 1: number analyzed (Participants) | 22 | 14
  First Intervention: Hour 1 | 16.10723481 [12.40927173 to 20.9071909] | 19.25708144 [13.98618037 to 26.51440036]
  First Intervention: Hour 4: number analyzed (Participants) | 22 | 15
  First Intervention: Hour 4 | 14.79254257 [11.76126752 to 18.60507937] | 16.80523147 [12.85367235 to 21.97160447]
  First Intervention: Hour 12: number analyzed (Participants) | 22 | 15
  First Intervention: Hour 12 | 17.06208571 [13.03988505 to 22.32494901] | 16.42411116 [11.98559242 to 22.50630741]

5. Secondary Outcome: Change in Oxygenation: Second Intervention
Description: The Oxygenation Index after the second intervention (if applicable) is calculated as the fraction of inspired oxygen, in percent, times the mean airway pressure, in mmHg, divided by the partial pressure of oxygen in arterial blood, in mmHg. Lower values are better.
Time Frame: 48 hours after enrollment, up to 12 hours after each intervention
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: index number
Arm/Group | Calfactant | Placebo (Air)
Number analyzed (Participants) | 16 | 14
index number
  Second Intervention: Hour 0: number analyzed (Participants) | 14 | 13
  Second Intervention: Hour 0 | 15.65261779 [10.74981818 to 22.79149651] | 15.05105738 [10.19615508 to 22.21762286]
  Second Intervention: Hour 1: number analyzed (Participants) | 15 | 12
  Second Intervention: Hour 1 | 21.28116857 [15.40809906 to 29.39286242] | 14.68059885 [10.36992308 to 20.78318046]
  Second Intervention: Hour 4: number analyzed (Participants) | 15 | 12
  Second Intervention: Hour 4 | 17.47108142 [13.41337922 to 22.75628541] | 15.40251337 [11.60739802 to 20.43846672]
  Second Intervention: Hour 12: number analyzed (Participants) | 14 | 12
  Second Intervention: Hour 12 | 17.26865232 [12.65514101 to 23.56404822] | 14.83842164 [10.66746181 to 20.64021983]

ADVERSE EVENTS:
Arm/Group | Calfactant | Placebo (Air)
All-Cause Mortality (participants affected / at risk) | 15/26 | 7/17
Serious Adverse Events (participants affected / at risk) | 15/26 | 7/17
Other Adverse Events (participants affected / at risk) | 8/26 | 1/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calfactant (N=26) | Placebo (Air) (N=17)
Death (Blood and lymphatic system disorders) | 15 (15) | 7 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Renal Failure (Renal and urinary disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Calfactant (N=26) | Placebo (Air) (N=17)
Peri-dosing hypotension (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Peri-dosing Hypoxia or Hypotension (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pneumomediatinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No